CLINICAL TRIAL: NCT05267483
Title: Evaluation of Usage Patterns and Outcomes in Patients Receiving Ceftolozane/Tazobactan (C/T) in Brazilian Hospitals
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: 15054519.3.0000.5249
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Sepsis
Keywords: Multidrug-Resistant (MDR) Bacterial Infections; Intensive Care Unit; Antibiotics; Ceftolozane/Tazobactan
MeSH Terms: conditions — Sepsis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Ceftolozane/Tazobactan (C/T) is a recent option to manage multidrug resistant gram-negative infections in hospital patients. Despite several randomized controlled trials describing safety and efficacy of C/T, real world evidence of its use, including indications, length of treatment and outcomes are lacking.

Understanding prescribing patterns of a new drug may help identifying possible knowledge gaps to target future randomized controlled trials. Additionally, real world evidence may help identifying practices and outcomes outside a clinical trial context.

DETAILED DESCRIPTION:
A multicenter, retrospective real-world study of hospitalized patients in a large private network of hospitals in Brazil (Rede D´Or São Luiz). Clinical data will be collected from Epimed Monitor Database®, an intensive care unit quality improvement database, which is in use over 1500 ICU beds, providing structured information on demographic, administrative and physiological parameters, as well as detailed data regarding the use of intensive care unit resources, infectious episodes, adverse events and checklists for adherence to best clinical practices. The pharmacy data is integrated from all hospitals in a single database, including clinical dosage, dosage form, route, dose regimen, duration of therapy. All sites are linked to a central microbiology lab with automatized systems and central online data. Data from Epimed®, pharmacist and business intelligence databases will be merged and medical records will be reviewed for the following information, which will be entered in a dedicated RedCap® form.

Indication for C/T as well as dosage, type of infusion and duration will be reviewed by a pharmacist and an infectious disease specialist. Reason for ceftolozane/tazobactam use was identified via medical record: physician notes, prescription changes and culture results.

Adverse events will be evaluated by an experienced pharmacist using a validated methodology (Naranjo algorithm).

Patient and infection outcome are classified as successful or failure at the end of the follow-up period. Patient outcome include ICU mortality and hospital 30-d mortality. A successful clinical infection resolution is defined as complete resolution of clinical signs and symptoms related to the infection treated by C/T and lack of microbiological evidence of infection. Clinical failure was defined as either lack of clinical response and/or recurrence and/or attributable mortality due to the infection. Outcomes will be stratified by C/T indication reason: initial empiric therapy, target therapy and failure of prior antibiotic therapy.

Cultures, identification of the organisms and susceptibility testing are performed at each participating center according to their own practice or by the central microbiology lab. The isolates are identified in genus and species by the VITEK® MS MALDI-TOF (bioMérieux - France) mass spectrometry methodology, and sensitivity and resistance criteria is defined using recent CLSI MIC breakpoints - M100, 28th Ed (Clinical and Laboratory Standards Institute - 2019).

ELIGIBILITY:
Inclusion Criteria:

1. aged > 18 years
2. received at least 2 days of C/T (with or without other antibiotics).

Exclusion Criteria:

1) Patients who were not hospitalized in the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in a large private network of hospitals in Brazil with severe infections, receiving ceftolozane/tazobactam for the treatment of proven or suspected infections.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Successful clinical infection resolution | 30 days
  Complete resolution of clinical signs and symptoms related to the infection treated by C/T and lack of microbiological evidence of infection
Clinical failure | 30 Days
  Defined as either lack of clinical response and/or recurrence and/or attributable mortality due to the infection.

SECONDARY OUTCOMES:
ICU mortality and hospital 30-d mortality | 30 days
  30 Days hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bozza, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Brazil